CLINICAL TRIAL: NCT03544541
Title: Association Between Metabolic Control and Cardiometabolic Risk in Children With Type 1 Diabetes.
Brief Title: Cardiometabolic Risk in Children With Type 1 Diabetes.
Status: Completed | Type: Observational
Sponsor: University of Ljubljana, Faculty of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: Cardio-Risk-T1D-SI
Record Dates: First submitted 2018-02-27; First posted 2018-06-01 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2019-11

CONDITIONS: Type1 Diabetes Mellitus; Metabolic Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To access the relationship between metabolic control of children and adolescents with type 1 diabetes and cardiometabolic risk through noninvasive imaging modalities to assess the early vasculature changes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for more than 0.5 year
* Age ≥ 10 years up to 25 years (inclusive)
* The subject/carer is willing to follow study specific instructions

Exclusion Criteria:

* Youth with maturity-onset diabetes of the young, hybrid, other, or missing type
* Any significant diseases / conditions including psychiatric disorders and substance abuse that in the opinion of the investigator is likely to affect the subject's ability to complete the study
* Current use of the following medications: medications that are used to lower blood glucose such as Pramlintide, Metformin and GLP-1 analogs. Beta blockers, glucocorticoids and other medications, which in the judgment of the investigator would be a contraindication to participation in the study (Anticoagulant therapy e.g. Plavix, LMW heparin, Coumadin, Immunosuppressant therapy)

Ages: 10 Years to 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: Nationwide cohort of children and adolescents with type 1 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Carotid Intima-Media Thickness | 24 months
  Non-invasive (Doppler Ultrasound) measurement of Carotid Intima-Media Thickness

CONTACTS AND LOCATIONS:
Locations (1):
- UMC-University Children's Hospital, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided